CLINICAL TRIAL: NCT00634387
Title: Effects of Anthocyans on Cardiovascular and Sympathetic Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: MedPalett (Unknown)
Responsible Party: Morten Rostrup MD PhD, Ullevaal University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC2008
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2010-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Anthocyans
  Interventions: Dietary Supplement: Anthocyans
- B (Placebo Comparator): no effective agent
  Interventions: Dietary Supplement: Anthocyans; Other: placebo

INTERVENTIONS:
Dietary Supplement: Anthocyans — Anthocyans
Other: placebo
  Arms: B
Dietary Supplement: Anthocyans
  Arms: A

SUMMARY:
Anthocyans modify cardiovascular and sympathetic function

ELIGIBILITY:
Inclusion Criteria:

* Ages 35 to 50 years old
* Males
* Hypertension

Ages: 35 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2008-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Systolic bloodpressure and heartrate

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular and Renal Research Center, Ulleval University Hospital, Oslo, Norway